CLINICAL TRIAL: NCT03091075
Title: Ability of Oral Steroid (Oxandrolone) to Halt Fatty Infiltration and Aid Rotator Cuff Healing: A Double-Blind, Randomized Clinical Trial
Brief Title: Oxandrolone Rotator Cuff Trial
Acronym: ORCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, George F. Hatch, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-17-00272
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Rotator Cuff; Anabolic Steroid; Testosterone; Oxandrolone
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Oxandrolone

STUDY DESIGN:
Intervention Model Description: Men and women aged 40 - 75 scheduled for rotator cuff repair, who have failed nonoperative management of chronic, full thickness rotator cuff tears confirmed by MRI, will be randomized into one of two groups, a control group (receiving placebo medication) and an experimental group receiving oral Oxandrolone for 12 weeks postoperative.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation will be performed using computer software and will occur at the pharmacy to ensure that all investigators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Oxandrolone
  Interventions: Drug: Oxandrolone
- Placebo Group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxandrolone — Treatment group will receive Oxandrolone daily for 12 weeks postoperatively
  Arms: Treatment Group
Drug: Placebo — Placebo group will receive placebo for 12 weeks postoperative
  Arms: Placebo Group

SUMMARY:
This study is about healing after a rotator cuff tear repair procedure. We hope to learn if a biologic medication: Oxandrolone, a synthetic derivative of the human hormone Testosterone (the principal male sex hormone and an anabolic steroid), given for 12 weeks following rotator cuff repair, is effective in aiding in the healing process and restoring muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for rotator cuff repair
* failed nonoperative management of chronic, full thickness rotator cuff tears
* full thickness rotator cuff tear confirmed on MRI

Exclusion Criteria:

* patients with prior shoulder surgery or prior rotator cuff repair
* tears larger than 5 cm
* significant glenohumeral arthritis (Hamada Grade 2 or higher)
* Untreated diabetes mellitus
* Pituitary tumor
* Rheumatoid arthritis
* Uncontrolled hypertension
* Congestive heart failure
* Myocardial infarction within the past 6 months
* End-stage renal disease
* Liver enzymes two times the normal value
* Deep Vein Thrombosis (DVT) within the past 6 months
* Disorder of the coagulation system
* Currently taking anticoagulation
* Claustrophobia
* Prior or current use of anabolic steroids
* Chromosomal disorders
* Prostate cancer
* Breast cancer
* Hypercalcemia
* Medications that interfere with testosterone production or function, including but not limited to 5 alpha-reductase inhibitors
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit through 6 weeks after the last dose of study treatment
* Any other condition or treatment interfering with completion of the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in structural integrity of the rotator cuff/tendon healing | baseline to 52 weeks
  assessed by MRI, classified based on the Sugaya classification and Goutallier Grade

SECONDARY OUTCOMES:
change in ASES shoulder score | baseline to 104 weeks
  American Shoulder Elbow Surgeon's Shoulder Score, Patient Questionnaire

OTHER OUTCOMES:
change in VAS pain scale | baseline to 104 weeks
  Visual Analog Score - pain scale, patient questionnaire
change in PASS Score | baseline to 104 weeks
  Patient Acceptable Symptom State, patient questionnaire
change in Functional Outcome - Shoulder Strength | baseline to 104 weeks
  isometric shoulder strength measures using a handheld dynamometer
change in Body Composition | baseline to 104 weeks
  body composition testing by bioelectric impedence

CONTACTS AND LOCATIONS:
Overall Officials: George R Hatch, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf SE, Thomas SJ, Dasu MR, Ferrando AA, Chinkes DL, Wolfe RR, Herndon DN. Improved net protein balance, lean mass, and gene expression changes with oxandrolone treatment in the severely burned. Ann Surg. 2003 Jun;237(6):801-10; discussion 810-1. doi: 10.1097/01.SLA.0000071562.12637.3E. PMID 12796576
- [Background] Jeschke MG, Finnerty CC, Suman OE, Kulp G, Mlcak RP, Herndon DN. The effect of oxandrolone on the endocrinologic, inflammatory, and hypermetabolic responses during the acute phase postburn. Ann Surg. 2007 Sep;246(3):351-60; discussion 360-2. doi: 10.1097/SLA.0b013e318146980e. PMID 17717439
- [Background] Schroeder ET, Vallejo AF, Zheng L, Stewart Y, Flores C, Nakao S, Martinez C, Sattler FR. Six-week improvements in muscle mass and strength during androgen therapy in older men. J Gerontol A Biol Sci Med Sci. 2005 Dec;60(12):1586-92. doi: 10.1093/gerona/60.12.1586. PMID 16424293
- [Background] Gerber C, Fuchs B, Hodler J. The results of repair of massive tears of the rotator cuff. J Bone Joint Surg Am. 2000 Apr;82(4):505-15. doi: 10.2106/00004623-200004000-00006. PMID 10761941
- [Background] Meyer DC, Wieser K, Farshad M, Gerber C. Retraction of supraspinatus muscle and tendon as predictors of success of rotator cuff repair. Am J Sports Med. 2012 Oct;40(10):2242-7. doi: 10.1177/0363546512457587. Epub 2012 Aug 27. PMID 22926748
- [Background] Sugaya H, Maeda K, Matsuki K, Moriishi J. Repair integrity and functional outcome after arthroscopic double-row rotator cuff repair. A prospective outcome study. J Bone Joint Surg Am. 2007 May;89(5):953-60. doi: 10.2106/JBJS.F.00512. PMID 17473131
- [Background] Goutallier D, Postel JM, Bernageau J, Lavau L, Voisin MC. Fatty muscle degeneration in cuff ruptures. Pre- and postoperative evaluation by CT scan. Clin Orthop Relat Res. 1994 Jul;(304):78-83. PMID 8020238
- [Background] Le BT, Wu XL, Lam PH, Murrell GA. Factors predicting rotator cuff retears: an analysis of 1000 consecutive rotator cuff repairs. Am J Sports Med. 2014 May;42(5):1134-42. doi: 10.1177/0363546514525336. Epub 2014 Apr 18. PMID 24748610
- [Background] Kim HM, Caldwell JM, Buza JA, Fink LA, Ahmad CS, Bigliani LU, Levine WN. Factors affecting satisfaction and shoulder function in patients with a recurrent rotator cuff tear. J Bone Joint Surg Am. 2014 Jan 15;96(2):106-12. doi: 10.2106/JBJS.L.01649. PMID 24430409
- [Background] Kelly BT, Kadrmas WR, Speer KP. The manual muscle examination for rotator cuff strength. An electromyographic investigation. Am J Sports Med. 1996 Sep-Oct;24(5):581-8. doi: 10.1177/036354659602400504. PMID 8883676
- [Background] Makhni EC, Steinhaus ME, Morrow ZS, Jobin CM, Verma NN, Cole BJ, Bach BR Jr. Outcomes assessment in rotator cuff pathology: what are we measuring? J Shoulder Elbow Surg. 2015 Dec;24(12):2008-15. doi: 10.1016/j.jse.2015.08.007. Epub 2015 Oct 21. PMID 26475640
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827
- [Background] Michener LA. Patient- and clinician-rated outcome measures for clinical decision making in rehabilitation. J Sport Rehabil. 2011 Feb;20(1):37-45. doi: 10.1123/jsr.20.1.37. PMID 21411821
- [Background] Mintken PE, McDevitt AW, Cleland JA, Boyles RE, Beardslee AR, Burns SA, Haberl MD, Hinrichs LA, Michener LA. Cervicothoracic Manual Therapy Plus Exercise Therapy Versus Exercise Therapy Alone in the Management of Individuals With Shoulder Pain: A Multicenter Randomized Controlled Trial. J Orthop Sports Phys Ther. 2016 Aug;46(8):617-28. doi: 10.2519/jospt.2016.6319. PMID 27477473
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Vitale MA, Vitale MG, Zivin JG, Braman JP, Bigliani LU, Flatow EL. Rotator cuff repair: an analysis of utility scores and cost-effectiveness. J Shoulder Elbow Surg. 2007 Mar-Apr;16(2):181-7. doi: 10.1016/j.jse.2006.06.013. PMID 17399623
- [Background] Ensor KL, Kwon YW, Dibeneditto MR, Zuckerman JD, Rokito AS. The rising incidence of rotator cuff repairs. J Shoulder Elbow Surg. 2013 Dec;22(12):1628-32. doi: 10.1016/j.jse.2013.01.006. Epub 2013 Mar 1. PMID 23466172
- [Background] Colvin AC, Egorova N, Harrison AK, Moskowitz A, Flatow EL. National trends in rotator cuff repair. J Bone Joint Surg Am. 2012 Feb 1;94(3):227-33. doi: 10.2106/JBJS.J.00739. PMID 22298054
- [Background] Lee TQ. Current biomechanical concepts for rotator cuff repair. Clin Orthop Surg. 2013 Jun;5(2):89-97. doi: 10.4055/cios.2013.5.2.89. Epub 2013 May 15. PMID 23730471
- [Background] Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40. doi: 10.2106/JBJS.D.02035. PMID 15930531
- [Background] Galatz LM, Ball CM, Teefey SA, Middleton WD, Yamaguchi K. The outcome and repair integrity of completely arthroscopically repaired large and massive rotator cuff tears. J Bone Joint Surg Am. 2004 Feb;86(2):219-24. doi: 10.2106/00004623-200402000-00002. PMID 14960664
- [Background] Bjornsson HC, Norlin R, Johansson K, Adolfsson LE. The influence of age, delay of repair, and tendon involvement in acute rotator cuff tears: structural and clinical outcomes after repair of 42 shoulders. Acta Orthop. 2011 Apr;82(2):187-92. doi: 10.3109/17453674.2011.566144. Epub 2011 Mar 24. PMID 21434791
- [Background] Moraiti C, Valle P, Maqdes A, Boughebri O, Dib C, Giakas G, Kany J, Elkholti K, Garret J, Katz D, Leclere FM, Valenti P. Comparison of functional gains after arthroscopic rotator cuff repair in patients over 70 years of age versus patients under 50 years of age: a prospective multicenter study. Arthroscopy. 2015 Feb;31(2):184-90. doi: 10.1016/j.arthro.2014.08.020. Epub 2014 Nov 11. PMID 25442647
- [Background] Gerber C, Meyer DC, Schneeberger AG, Hoppeler H, von Rechenberg B. Effect of tendon release and delayed repair on the structure of the muscles of the rotator cuff: an experimental study in sheep. J Bone Joint Surg Am. 2004 Sep;86(9):1973-82. doi: 10.2106/00004623-200409000-00016. PMID 15342760
- [Background] Patel S, Gualtieri AP, Lu HH, Levine WN. Advances in biologic augmentation for rotator cuff repair. Ann N Y Acad Sci. 2016 Nov;1383(1):97-114. doi: 10.1111/nyas.13267. Epub 2016 Oct 17. PMID 27750374
- [Background] Ruiz-Moneo P, Molano-Munoz J, Prieto E, Algorta J. Plasma rich in growth factors in arthroscopic rotator cuff repair: a randomized, double-blind, controlled clinical trial. Arthroscopy. 2013 Jan;29(1):2-9. doi: 10.1016/j.arthro.2012.08.014. PMID 23276410
- [Background] Rodeo SA, Delos D, Williams RJ, Adler RS, Pearle A, Warren RF. The effect of platelet-rich fibrin matrix on rotator cuff tendon healing: a prospective, randomized clinical study. Am J Sports Med. 2012 Jun;40(6):1234-41. doi: 10.1177/0363546512442924. Epub 2012 Apr 10. PMID 22495146
- [Background] Gulotta LV, Kovacevic D, Ehteshami JR, Dagher E, Packer JD, Rodeo SA. Application of bone marrow-derived mesenchymal stem cells in a rotator cuff repair model. Am J Sports Med. 2009 Nov;37(11):2126-33. doi: 10.1177/0363546509339582. Epub 2009 Aug 14. PMID 19684297
- [Background] Gerber C, Meyer DC, Nuss KM, Farshad M. Anabolic steroids reduce muscle damage caused by rotator cuff tendon release in an experimental study in rabbits. J Bone Joint Surg Am. 2011 Dec 7;93(23):2189-95. doi: 10.2106/JBJS.J.01589. PMID 22159854
- [Background] Gerber C, Meyer DC, Fluck M, Benn MC, von Rechenberg B, Wieser K. Anabolic Steroids Reduce Muscle Degeneration Associated With Rotator Cuff Tendon Release in Sheep. Am J Sports Med. 2015 Oct;43(10):2393-400. doi: 10.1177/0363546515596411. Epub 2015 Aug 24. PMID 26304962
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03091075/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03091075/ICF_001.pdf